CLINICAL TRIAL: NCT05413564
Title: Impact of a Self-Exclusion Procedure Optimized by an Extension of the Suspension of Commercial Solicitations
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: LOCAL 2021 /AL
Record Dates: First submitted 2022-05-24; First posted 2022-06-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimized self-exclusion procedure A (Other): optimized self-exclusion procedure by extending the suspension of commercial solicitations for a total of 9 months
  Interventions: Other: optimized self-exclusion procedure by extending the suspension of commercial solicitations for a total of 9 months
- standard procedure (Other): standard self-exclusion procedure B
  Interventions: Other: optimized self-exclusion procedure by extending the suspension of commercial solicitations for a total of 9 months

INTERVENTIONS:
Other: optimized self-exclusion procedure by extending the suspension of commercial solicitations for a total of 9 months — optimized self-exclusion procedure A

SUMMARY:
Considering that self-exclusion from gambling on a particular website is an intervention for and by individuals who have developed a gambling disorder, it is currently exclusively a behavioural intervention in the sense that it prevents the behaviour Resumption of commercial solicitations only in the period when gambling is not accessible in the corresponding website , through voluntary self-exclusion (where the gambler prevents himself or herself from gambling), does not appear to be sufficient to prevent relapse. Early commercial solicitations, in the immediate intercourse after the end of the self-exlcusion period may precipitate relapse in gamblers whose behaviour change is by definition recent, and who have only received a behavioural measure. The investigators hypothesize an improved efficacy as measured by reduced gambling after a self-exclusion optimized by a period of suspension of commercial solicitations extended to 9 months, compared to self-exclusion with the standard procedure. Gamblers will be randomized according to an a priori randomization list.

DETAILED DESCRIPTION:
This is a study evaluating the impact of PMU's implementation of an optimized self-exclusion procedure by extending the suspension of commercial solicitations for a total of 9 months, the self-exclusion being referred to as a non-medical "responsible gambling" tool, compared to the standard procedure. The self-excluded gamblers will be randomized according to an a priori randomization list, and will receive either the optimized self-exclusion procedure A or the standard self-exclusion procedure B. The study consists of a comparison between two groups A and B. The study involves non-medical gambling and socio-demographic data, routinely recorded in a regulatory manner with a permanent CNIL authorization PMU.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* self-excluder during the recruitment period
* Online sports betting
* poker and horse racing player
* account opened for at least 4 weeks
* self-exclusion for 3 months or less (minimum 3 days).

Exclusion Criteria:

* Player who has objected to the use of his collected data when opening his account.
* It's not the first self-exclusion of the inclusion period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2554 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
change in total net loss | over the last 4 weeks,between the last 4 weeks before self-exclusion T0, and the last 4 weeks at 9 months T2
  Evaluate the effect of the self-exclusion procedure optimized by extending the suspension of commercial solicitations for a total of 9 months, compared to the existing procedure, on the intensity of gambling.

SECONDARY OUTCOMES:
change in total net loss | between last 4 weeks prior to self-exclusion, and last 4 weeks at 6 months T1, 12 months T3 and 18 months T4
  Evaluate early efficacy at 6 months, maintenance of efficacy at 18 months comparison of changes according to type of play

CONTACTS AND LOCATIONS:
Locations (1):
- Amandine LUQUIENS, Nîmes, Nîmes, France

REFERENCES:
- [Derived] von Hammerstein C, Benyamina A, Luquiens A. Long-term efficacy of an optimized online gambling self-exclusion procedure with extended suspension of commercial solicitations: a randomized controlled trial. Harm Reduct J. 2025 Dec 30;22(1):204. doi: 10.1186/s12954-025-01339-0. PMID 41469674